CLINICAL TRIAL: NCT01471093
Title: Safety Study of OPC-12759 Ophthalmic Solution in Healthy Subjects
Brief Title: Safety Study of OPC-12759 Ophthalmic Solution
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 037E-11-004; JapicCTI-111674 (Other: Japic)
Record Dates: First submitted 2011-11-03; First posted 2011-11-11 (Estimated); Results first posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Solution (Experimental): A single dose of OPC-12759 Ophthalmic solution for two-day treatment
  Interventions: Drug: OPC-12759 Ophthalmic solution
- Suspension (Active Comparator): A single dose of OPC-12759 Ophthalmic suspension for two-day treatment
  Interventions: Drug: OPC-12759 Ophthalmic suspension

INTERVENTIONS:
Drug: OPC-12759 Ophthalmic solution — 2％ OPC-12759 Ophthalmic solution
  Arms: Solution
Drug: OPC-12759 Ophthalmic suspension — 2％ OPC-12759 Ophthalmic suspension
  Arms: Suspension

SUMMARY:
The purpose of this study is to assess the safety of OPC-12759 ophthalmic solution in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* BMI : {body weight (kg) / [height (m)] 2 } must be 17.6 or greater, and less than 26.4 kg/m2

Exclusion Criteria:

1. Presence of ocular disorder
2. Intraocular pressure of 21mmHg or higher
3. Corrected visual acuity of less than 1.0
4. Dysfunction of nasolacrimal duct or history of surgery related to nasolacrimal duct or eye lid which affects the nasolacrimal outflow
5. History of refractive surgery
6. History of other ocular surgeries within 12 months
7. Those who cannot discontinue the use of contact lenses from the 1st dose to 5-hour-post-dose

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-11; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eiji Murakami, Study Chair — Director of Division of Dermatologicals and Ophthalmologicals, Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Kansai region, Osaka, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a single-center, randomized, crossover, open-label study.
Groups:
- OPC-12759 Solution With Nasal Root Pressed, Then OPC-12759 Solution Without Nasal Root Pressed; OPC-12759 Solution Without Nasal Root Pressed, Then OPC-12759 With Nasal Root Pressed: One drop of 2% OPC-12759 ophthalmic solution was instilled into each eye once. Subjects who were instructed to press the nasal root at the first instillation (n=25) were asked not to press it at the second instillation, and subjects who were instructed not to press the nasal root at the first instillation (n=25) were asked to press it at the second instillation.
  The second instillation was conducted within 14 days after the first instillation.
- OPC-12759 Suspension With Nasal Root Pressed, Then OPC-12759 Solution Without Nasal Root Pressed; OPC-12759 Suspension Without Nasal Root Pressed, Then OPC-12759 Solution With Nasal Root Pressed: One drop of OPC-12759 ophthalmic suspension was instilled into each eye once. Subjects who were instructed to press the nasal root at the first instillation (n=25) were asked not to press it at the second instillation, and subjects who were instructed not to press the nasal root at the first instillation (n=25) were asked to press it at the second instillation.
  The second instillation was conducted within 14 days after the first instillation.
Period: Overall Study
Arm/Group | OPC-12759 Solution With Nasal Root Pressed, Then OPC-12759 Solution Without Nasal Root Pressed | OPC-12759 Solution Without Nasal Root Pressed, Then OPC-12759 With Nasal Root Pressed | OPC-12759 Suspension With Nasal Root Pressed, Then OPC-12759 Solution Without Nasal Root Pressed | OPC-12759 Suspension Without Nasal Root Pressed, Then OPC-12759 Solution With Nasal Root Pressed
Started | 25 | 25 | 25 | 25
Completed | 24 | 25 | 25 | 25
Not Completed | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- OPC-12759 Solution: One drop of 2% OPC-12759 ophthalmic solution was instilled into each eye once.
- OPC-12759 Suspension: One drop of OPC-12759 ophthalmic suspension was instilled into each eye once.
- Total: Total of all reporting groups
Arm/Group | OPC-12759 Solution | OPC-12759 Suspension | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.8 (6.3) | 25.9 (6.3) | 26.9 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 27 | 55
  Male | 22 | 23 | 45
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Blurred Vision After Instillation
Description: The number of subjects with white blurred vision after first and/or second instillation was calculated for subjects.
Time Frame: The first and second instillation
Population: Analysis set consisted of all subjects who had received the investigational product at least once.
Measure: Number; unit: participants
Groups:
- OPC-12759 Solution With Nasal Root Pressed/Not Pressed: One drop of 2% OPC-12759 ophthalmic solution was instilled into each eye once. Subjects who were instructed to press the nasal root at the first instillation (n=25) were asked not to press it at the second instillation, and subjects who were instructed not to press the nasal root at the first instillation (n=25) were asked to press it at the second instillation.
  The second instillation was conducted within 14 days after the first instillation.
- OPC-12759 Suspension With Nasal Root Pressed/Not Pressed: One drop of OPC-12759 ophthalmic suspension was instilled into each eye once. Subjects who were instructed to press the nasal root at the first instillation (n=25) were asked not to press it at the second instillation, and subjects who were instructed not to press the nasal root at the first instillation (n=25) were asked to press it at the second instillation.
  The second instillation was conducted within 14 days after the first instillation.
Arm/Group | OPC-12759 Solution With Nasal Root Pressed/Not Pressed | OPC-12759 Suspension With Nasal Root Pressed/Not Pressed
Number analyzed (Participants) | 50 | 50
participants
  With Nasal Root Press | 0 | 10
  Without Nasal Root Press: number analyzed (Participants) | 49 | 50
  Without Nasal Root Press | 0 | 21

2. Primary Outcome: Number of Subjects With Bitter Taste
Description: The number of subjects with bitter taste on first and/or second instillation was calculated for subjects.
Time Frame: The first and second instillation
Population: Analysis set consisted of all subjects who had received the investigational product at least once.
Measure: Number; unit: participants
Arm/Group | OPC-12759 Solution With Nasal Root Pressed/Not Pressed | OPC-12759 Suspension With Nasal Root Pressed/Not Pressed
Number analyzed (Participants) | 50 | 50
participants
  With Nasal Root Press | 33 | 23
  Without Nasal Root Press: number analyzed (Participants) | 49 | 50
  Without Nasal Root Press | 41 | 29

ADVERSE EVENTS:
Time Frame: Treatment period (2 days up to 15 days)
Description: Safety analysis set consisted of all subjects who had received the investigational product at least once.
  White blurred vision after instillation and bitter taste were not considered to be adverse events because they were the specific symptoms for study evaluation.
  Adverse Events detected were systemic and not attributable to one specific intervention or another.
Groups:
- OPC-12759 Solution: One drop of 2% OPC-12759 ophthalmic solution was instilled into each eye (instillation was conducted twice, the second instillation was within 14 days after the first instillation).
- OPC-12759 Suspension: One drop of OPC-12759 ophthalmic suspension was instilled into each eye (instillation was conducted twice, the second instillation was within 14 days after the first instillation).
Arm/Group | OPC-12759 Solution | OPC-12759 Suspension
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 6/50 | 2/50
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OPC-12759 Solution (N=50) | OPC-12759 Suspension (N=50)
Chalazion (Eye disorders) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Protein urine present (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No